CLINICAL TRIAL: NCT06697756
Title: The Effect of Manipulating the Perception of Effort During Resistance Exercise Training on Glycemic Control and Psychological Responses in Individuals Living With Prediabetes: a Randomized-controlled Trial
Brief Title: Resistance Training for the Improvement of Glycemic Control in Prediabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Flavio de Castro Magalhaes, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2409157184
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Prediabetes (Insulin Resistance, Impaired Glucose Tolerance)
Keywords: resistance training; glycemic control
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: Participants will undergo anthropometrics, familiarization, and strength test, and will be randomized to a high-effort, or a low-effort resistance training protocol, that will be carried out 2 days/week, for 16 weeks, and will be composed of 7 exercises (hex bar squat, seated chest press, leg press, lat pulldown, leg extension, shoulder press, leg curl, always in this order). Load will be set at 10-RM load (75% 1-RM). Participants will be instructed to perform the concentric (lifting) phase of the repetition as fast as they can (~0.5 seconds), and to perform the eccentric phase in 2 seconds. Psychological responses (perceived exertion, enjoyment, feeling scale, discomfort, and self-efficacy) will be assessed. Anthropometrics will be repeated after training, and before and after the training period, glycemic control will be assessed via a continuous glucose monitoring device. The main outcomes will be compared between training interventions, pre-training data will used as comparator.
Who Masked: Outcomes Assessor
Masking Description: Data and statistical analysis will be performed by a researcher blinded to groups and participants' identities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-effort (Experimental): The high-effort protocol will entail performing 3 sets per exercise, 8 repetitions per set, ~2.5 seconds per repetition, with 120 seconds between sets and exercises.
  Interventions: Behavioral: High-effort resistance exercise training
- Low-effort (Experimental): The low-effort protocol will entail performing 6 sets per exercise, 4 repetitions per set, ~2.5 seconds per repetition, with 60 seconds between sets and exercises.
  Interventions: Behavioral: Low-effort resistance exercise training

INTERVENTIONS:
Behavioral: High-effort resistance exercise training — Six sets per exercise, 8 repetitions per set.
  Arms: High-effort
Behavioral: Low-effort resistance exercise training — Three sets per exercise, 4 repetitions per set.
  Arms: Low-effort

SUMMARY:
The purpose of this research is to study the effects of resistance exercise training with different degrees of effort on your glucose responses (what we call glycemic control) and psychological responses.

DETAILED DESCRIPTION:
Type 2 diabetes is a disease where peripheral insulin resistance associated with pancreatic beta-cell dysfunction leads to chronically elevated blood glucose levels. Type 2 diabetes is preceded by prediabetes, a condition where blood glucose levels are higher than normal, but not enough to be considered type 2 diabetes. One in 3 Americans 18 years-old or over is living with prediabetes and their risk of developing type 2 diabetes is ~50%. Importantly, prediabetes is a treatable condition, it has been shown that exercise interventions are more effective than metformin (the most commonly prescribed hypoglycemic oral mediation) for the improvement in glucose control in individuals living with prediabetes.

Although regular exercise is highly recommended for the management and improvement of glycemic control for individuals living with prediabetes, adherence to exercise interventions is lower than those without prediabetes. The reasons individuals do not engage in regular exercise are multifaceted, but often relate to low self-efficacy (self-perception of the ability to accomplish something), and perceiving exercise as uncomfortable. In fact, those factors have been shown to predict exercise behavior in individuals living with prediabetes and type 2 diabetes. Thus, strategies aiming at improving feelings and perceptions during exercise, while retaining the positive improvement on glucose metabolism, can potentially increase long-term exercise adherence for individuals living with prediabetes.

Aerobic exercise is usually the default exercise prescribed for individuals living with prediabetes. However, as most individuals living with prediabetes are overweight and sedentary, even a brisk walk can be difficult, uncomfortable or painful, and resistance exercise training can be a more attractive and easier form of exercise. Moreover, there is vast literature showing that resistance exercise training improves glycemic control in individuals living with prediabetes and type 2 diabetes. Importantly, resistance exercise training has been shown to reduce prediabetes prevalence in individuals living with prediabetes. Altogether, resistance exercise training can be both effective for the prevention of type 2 diabetes and appealing for individuals living with prediabetes, and has been shown to be a viable exercise prescription option for this population. Not surprisingly, resistance exercise training prescription for individuals living with prediabetes and type 2 diabetes is widely recommended by international guidelines.

Resistance exercise training prescription entails the manipulation of many variables. These include exercise type (single- or multi-joint) and order, load, number of sets per exercise, repetitions per set, repetition duration (aka tempo), and resting interval between sets. There are also variables that are derived from the above, such as total volume-load (load x sets x reps), and session density (total volume-load divided by session duration). Appropriate manipulation of these variables is regarded as important for targeting specific adaptations. More recently, attention has also been directed to the degree of effort during resistance exercise training sets as a potentially important variable that can be manipulated to affect adaptative outcomes. In fact, it has been suggested that the degree of effort is important for improvements in glucose metabolism and insulin sensitivity in individuals living with type 2 diabetes, although direct evidence of that is lacking. However, performing resistance exercise sets with a high degree of effort is associated with higher perceived exertion and discomfort, increased muscle soreness, negative perceptual responses, and higher neuromuscular fatigue and muscle damage. Taken together, these negative perceptual and physiological responses to resistance exercise sets performed with high degree of effort might negatively affect enjoyment, self-efficacy, and motivation during a resistance exercise session, ultimately reducing long-term adherence. Individuals living with prediabetes might be even more susceptible to these negative responses, because as stated earlier, their physical activity levels are particularly low, and they identify lack of motivation and low self-efficacy as barriers for being more physically active.

Therefore, resistance exercise training prescriptions should to be tailored to meet not only the glycemic control needs of individuals living with prediabetes, but also their motivation and self-perceived capacity to engage in, and long-term adhere to exercise. Thus, the primary aim of this study is to assess the effects resistance exercise training with different degrees of effort on glycemic control and psychological responses in individuals living with prediabetes. Although the degree of effort has been suggested to play an important role in the beneficial effects of resistance exercise on glucose and insulin responses in individuals living with type 2 diabetes, this has not been tested directly, nor it is known if this also applies to individuals living with prediabetes. Also, perceptual responses will be assessed to investigate how feelings experienced during resistance exercise training are altered relative to different degrees of effort. The hypothesis is that glycemic control will not be affected by the degree of effort, and improvements will be observed regardless of that. Also, it is hypothesized that the low degree of effort will be associated with better psychological responses. As a secondary aim, adherence rate and reasons for adhering or not to the protocols will be thoroughly investigated and reported. It is anticipated that better adherence will be associated with the low degree of effort and psychological responses experienced during training.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years;
* presence of prediabetes (fasting glycemia between 100 and 125 mg/dL or glycated hemoglobin [A1c] between 5.7 and 6.4%).

Exclusion Criteria:

* Have a significant cognitive impairment,
* Are non-ambulatory,
* Have lower extremity amputation,
* Have renal failure,
* Have liver disease,
* Have uncontrolled hypertension (>160 mmHg systolic and/or >100 mmHg diastolic),
* Have unstable cardiovascular disease,
* Have a history of severe cardiovascular problems,
* Have decompensated heart failure,
* Have uncontrolled arrhythmias,
* Have severe pulmonary hypertension (mean pulmonary arterial pressure >55 mm Hg),
* Have severe and symptomatic aortic stenosis,
* Have acute myocarditis, endocarditis, or pericarditis,
* Have aortic dissection,
* Have Marfan syndrome,
* Have unrepaired aortic aneurysm,
* Have proliferative diabetic retinopathy,
* Have rapidly progressive terminal illness,
* Are unable to perform resistance exercise to due preexisting musculoskeletal conditions (e.g., joint pain, chronic injury or tendinopathy),
* Are under biguanide (metformin) treatment, but are taking for less than 3 months,
* Have taken drugs known to increase the risk of tendon disorders (e.g., tendinopathy and tendon rupture) within the last 6 months. These drugs include, but may not be limited to: fluoroquinolones, glucocorticoids, aromatase inhibitors, anabolic steroids, antiretrovirals, isotretinoin, cephalexin, rituximab, sitagliptin, cephalosporins, azithromycin, and sulfonamides.
* Are pregnant or trying to become pregnant during the study,
* Are prisoners,
* Are persons that require a legally authorized representative.

Temporary exclusions include:

* Being subjected to recent surgeries for which resistance training is not recommended,
* Have symptomatic hernias,
* Have acute illness,
* Have recent fractures, or other injuries until resolved.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Glucose concentration | For 60 hours before the first training session and for 60 hours after the last (32nd) training session
  Average glucose concentration (measured in milligrams per deciliter of blood, with a continuous glucose monitoring device)

SECONDARY OUTCOMES:
Adherence to the resistance training protocols | From date of randomization until the date of first documented dropout from any cause, assessed up to 16 weeks (the end of the training period)
  Adherence rate assessed using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Locations (1):
- UNM Exercise Physiology Lab, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
For sharing the data generated the Open Science Framework (OSF) platform will be used. Before data sharing, all personal identifiers will be stripped from the data. Specifically, any direct identifiers (e.g., name, email addresses, phone and cell phone numbers), date identifiers (e.g., birthday, date of disease diagnosis, dates patients participated in data collection), location identifiers (e.g., personal or professional addresses, zip codes), links to external datasets identifiers (e.g., social media accounts) will be removed. Furthermore, participants will be represented by an identification string generated randomly (www.random.org/strings/), and their data will be inserted in the files in a random order, not associated with the order they were enrolled. Thus, data will be entirely de-identified before sharing, in order to protect sensitive personal information and privacy.
Time Frame: The anticipated date for data sharing will be 6 months after publication of data or 18 months after award end date, whatever happens first.
Access Criteria: Open access